CLINICAL TRIAL: NCT07306416
Title: Acute Effects of Tissue Flossing on the Viscoelastic Properties of the Muscles and Jump Performance in Handball Players: a Crossover Design
Brief Title: Acute Effects of Tissue Flossing on Muscle Properties and Jump Performance in Handball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 177/2020
Record Dates: First submitted 2025-08-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-08

CONDITIONS: Tissue Flossing
Keywords: Myofascial Release Therapy; Tissue Flossing; Foam rolling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tissue Flossing conditioning (Experimental): Tissue flossing using a 5 cm x 3.5 m green Sanctband Comprefloss band was wrapped around the thigh area. After the floss band was applied, the participants did 10 bodyweight squats, making sure to bend their knees to a 90-degree angle. Next, they did 10 dynamic lunges on each leg, switching legs after each lunge. After finishing these exercises, the floss band was removed.
  Interventions: Other: Tissue Flossing conditioning
- Foam rolling conditioning (Experimental): Each participant rolled the quadriceps on the right, then the left, for 30 seconds each, and did the same for the hamstrings, starting with the right and then the left, also for 30 seconds each side.
  Interventions: Other: Foam Rolling
- No intervention (No Intervention): Participants perform standard dynamic warm-up exercises (bodyweight squats and lunges) with no additional device or treatment.

INTERVENTIONS:
Other: Tissue Flossing conditioning — Tissue flossing using a 5 cm x 3.5 m green Sanctband Comprefloss band was wrapped around the thigh area. After the floss band was applied, the participants did 10 bodyweight squats, making sure to bend their knees to a 90-degree angle. Next, they did 10 dynamic lunges on each leg, switching legs after each lunge. After finishing these exercises, the floss band was removed.
  Arms: Tissue Flossing conditioning
Other: Foam Rolling — Using a firm foam roller to roll the quadriceps and hamstrings for 30 seconds per side.
  Arms: Foam rolling conditioning

SUMMARY:
Purpose of the Study This study looked at how two popular warm-up techniques-tissue flossing and foam rolling-affect muscle flexibility, muscle properties, and jumping ability in young male handball players. The goal was to see which method might be better for preparing athletes for performance.

What Are These Techniques?

Tissue flossing: Wrapping a special elastic band tightly around a muscle or joint for a short time while moving. This temporarily reduces blood flow, and when the band is removed, blood rushes back in, which may boost muscle readiness.

Foam rolling: Using your body weight to roll muscles over a firm foam cylinder. This applies pressure to the muscle and fascia, helping to relax tight areas and increase flexibility.

Who Took Part? 30 male handball players, around 17 years old, who were healthy and injury-free. None had regularly used tissue flossing or foam rolling before.

How Was the Study Done?

Each player tried all three conditions on separate days:

Tissue flossing

Foam rolling

Control (no special technique, just exercises)

Before and after each session, the researchers measured:

Active range of motion (AROM) - how far they could move their leg muscles without help

Muscle properties - stiffness and tone of key thigh muscles

Jump performance - height and speed of force production in a countermovement jump

Measurements were taken before, 2 minutes after, and 15 minutes after each warm-up.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified male
* Aged approximately 16-18 years
* Active handball player with at least 8 years of playing experience
* Currently healthy with no injuries in the past 3 months
* Able to perform physical activity and complete all testing procedures
* No prior regular use of tissue flossing (TF) or foam rolling (FR) techniques

Exclusion Criteria:

* Current or recent (within 3 months) musculoskeletal injury
* Any medical condition that would limit safe participation in exercise testing
* Previous experience with tissue flossing (TF) or regular use of foam rolling (FR)
* Inability to follow study instructions or complete all sessions

Ages: 15 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The study specifically recruited male handball players aged around 17 years, so this reflects the protocol accurately.
Enrollment: 30 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Active Range of Motion | Before the intervention, 2 minutes after, and 15 minutes after the intervention.
  Measured using the Active Knee Extension (AKE) test for both legs to assess hamstring flexibility.

SECONDARY OUTCOMES:
Jump Performance - Jump Height | Before the intervention, 2 minutes after, and 15 minutes after the intervention.
  Height achieved in a countermovement jump (CMJ) without arm swing, measured with a force plate.
Jump Performance - Braking Rate of Force Development | Before the intervention, 2 minutes after, and 15 minutes after the intervention.
  The rate at which force is developed during the braking phase of the CMJ, measured via force plate.

OTHER OUTCOMES:
Viscoelastic Muscle Properties - Stiffness | Before the intervention, 2 minutes after, and 15 minutes after the intervention.
  Muscle stiffness of the rectus femoris (RF), vastus lateralis (VL), and biceps femoris (BF) in both legs, measured with the MyotonPRO device
Viscoelastic Muscle Properties - Tone | Before the intervention, 2 minutes after, and 15 minutes after the intervention
  Muscle tone (oscillation frequency) of the RF, VL, and BF in both legs, measured with the MyotonPRO device.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Sport at Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article will be made available upon reasonable request to the corresponding author (anna.pisz@ftvs.cuni.cz). Data will be available immediately following publication, with no end date.
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2025-08-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT07306416/Prot_000.pdf